CLINICAL TRIAL: NCT01090830
Title: Phase Ib/II Study to Determine the Recommended Dose, Safety, and Preliminary Efficacy of Belinostat When Used in Combination With Carboplatin, Paclitaxel, and Bevacizumab in Patients With Untreated Non-small Cell Lung Cancer.
Brief Title: Safety and Efficacy of Belinostat When Used With Standard of Care Chemotherapy for Untreated Non-small Cell Lung Cancer
Acronym: HCH003
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Principal Investigator has left institution. IND withdrawn.
Sponsor: Holy Cross Hospital, Florida (Other)
Responsible Party: Principal Investigator, Paul Papagni, Executive Director of Clinical Research, Holy Cross Hospital, Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HCH003
Record Dates: First submitted 2010-03-22; First posted 2010-03-23 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2013-03

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non small cell lung cancer; Belinostat; carboplatin; Paclitaxel; Bevacizumab; chemotherapy; Maximum Tolerated Dose; Neoplasms, Pulmonary; Lung Cancer; Event Free Survival; Disease free survival; Progression Free Survival; Histone Deacetylase Inhibitors; Treatment Efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — belinostat; Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Belinostat (Experimental): This is a one arm, open label study of the investigational medication Belinostat.
  Interventions: Drug: Belinostat, carboplatin, paclitaxel and bevacizumab

INTERVENTIONS:
Drug: Belinostat, carboplatin, paclitaxel and bevacizumab — Induction therapy will include 6 cycles of 5-days of medication administration followed by a 16 day rest period. Belinostat will be given once a day for 5 days total. Three dose levels will be evaluated (600mg/kg, 800 mg/kg, and 1000 mg/kg). In addition, participants will receive fixed doses of intravenous carboplatin (AUC 6), Paclitaxel (200 mg/m2), and bevacizumab (15 mg/kg) once on day 3 of each cycle. Serial disease status evaluations will be done throughout the study.
  In the absence of significant toxicity or disease progression, participants may continue with a maintenance regimen of bevacizumab and Belinostat for an additional 6 cycles. The dose of Belinostat received during maintenance will be that tolerated in the initial 6 cycles.
  Other Names: Belionostat; PDX101; Bevacizumab; Carboplatin; Paraplatin; Paclitaxel; Taxol

SUMMARY:
The purpose of this study is to establish the safest dose of the investigational medication Belinostat that can be administered with a standard of care chemotherapy regimen of bevacizumab, carboplatin, and paclitaxel. Further study will examine the short and long-term effect (up to 2 years) of this medication on participant's disease status and overall survival.

DETAILED DESCRIPTION:
This is a Phase Ib/II, single center, open label, dose-finding study to evaluate the use of Belinostat when given with standard of care chemotherapy in patients with untreated, non-small cell lung cancer (NSCLC). In the Phase Ib portion, dose limiting toxicity evaluation will be used to determine the maximum tolerated dose (MTD) of Belinostat when given with fixed doses of bevacizumab, carboplatin, and paclitaxel(a BelCap-B regimen). Three dose levels of Belinostat are proposed (600mg/kg, 800mg/kg, 1000mg/kg). Determination of MTD will be the basis for establishing set dosing for the phase II component of the study.

The phase II portion of the study includes further drug safety evaluation and a preliminary assessment of efficacy of Belinostat when used with specified induction and maintenance regimens. Response will be evaluated through the RECIST criteria. Additional analysis will be done to estimate the time to response, progression free survival, median survival, and overall survival (OS) in study participants to 2 years post-initiation of cycle 1.

Based on a standard 3 x 3 statistical design, the phase Ib portion may accrue between 3 to 12 participants. Phase II will have a minimum sample size of 10 and a maximum of 16 patients. Participants who complete the Phase I portion and are able to advance to Phase II, will be evaluable for the Phase II objectives.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented NSCLC confirmed.
* Has advanced NSCLC (Stage IV), not previously treated with any chemotherapy regiment (prior adjuvant chemotherapy and/or chemotherapy/radiation for Stage III allowed).
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Life expectancy of > 3 months
* Must have returned to baseline or grade 1 adverse event from any acute toxicity related to prior therapy
* Adequate immune and multisystem organ function (as evidenced by urine and blood values within specified parameters).

Exclusion Criteria:

* Brain or meningeal metastases. Note, patients with adequately treated brain metastases, e.g. surgically resected, or adequately controlled by radiotherapy, with no residual neurological symptoms due to metastases and no steroid treatment required, can be enrolled. If clinical suspicion, adequate investigations should be performed to rule out brain metastases or meningeal involvement.
* History of a previous malignancy within 5 years with the exception of non-metastatic non-melanoma skin cancer or cervical carcinoma in situ. Prior systemic therapy for other malignancy must be completed at least 5 years before treatment is allowed.
* Lung carcinoma of squamous cell histology (mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is not acceptable).
* History of hemoptysis within 3 months prior to enrollment
* Current or recent (within 10 days of enrollment) use of aspirin (>325 mg/day) or chronic use of other non-steroidal anti-inflammatory medications.
* Prior systemic anti-tumor therapy for Stage IV lung cancer. Note, prior radiotherapy is allowed provided treatment was completed at least 2 weeks before enrollment. Prior surgery is allowed if completed at least 4 weeks before enrollment.
* Treatment with investigational agents within the 2 weeks prior to enrollment.
* Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease.
* Hypertension not controlled by medical therapy.
* Significant cardiovascular disease, myocardial infarction within the past 6 months, unstable angina, unstable arrhythmia or a need for anti-arrhythmic therapy (use of medication to control heart rate in patients with atrial fibrillation is allowed, if stable medication for at least last month prior to enrollment, or evidence of acute ischemia on electrocardiogram).
* Marked baseline prolongation of QT/QTc interval that required use of concomitant medication that may cause Torsade de Pointes
* Significant, non-healing wounds, acute or non-healing ulcers, or bone fractures within 3 months of fracture.
* Undergone major surgery within 4 weeks of planned initiation of cycle 1.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of enrollment.
* History of any gastrointestinal bleeding within the 3 months prior to enrollment.
* Known hypersensitivity to either platinum compounds or paclitaxel, or any components of the study medications, and inability for desensitization.
* Peripheral neuropathy NCI ≥ Grade 2.
* Co-existing active severe infection or any co-existing medical condition likely to interfere with trial procedures.
* Known infection with HIV, or known active Hepatitis B or C infection.
* Pregnant or lactating.
* not willing to use effective contraception during the study and until 6 months post-completion of last cycle administered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The recommended phase II dose of Belinostat when used in combination with carboplatin, paclitaxel and bevacizumab. | 1 year
  The aim of the initial phase Ib component is to establish the maximum tolerated dose (MTD) of Belinostat when used with a standard of care carboplatin, paclitaxel and bevacizumab course of therapy ("BelCap-B") regimen. The MTD will be determined through the process of dose-limiting-toxicity evaluation.

SECONDARY OUTCOMES:
To evaluate overall survival with this investigational treatment. | 2 years
  The percentage of participants who are alive at 2 years post initiation of investigational treatment.
Long-term safety (late-effects up to 2 years) | 2 years
  Long-term (up to 2 years) safety evaluation of the investigational treatment will be evaluated by ongoing evaluation of adverse events/late-effects using the NCI Common Toxicity Criteria.
Evaluate disease response of participants who receive this investigational medication regimen | 2 years
  Response to therapy will be measured by the RECIST criteria. The investigators will assess the percentage of research participants whose disease status indicates a response to investigational treatment according to the RECIST criteria.
To evaluate progression-free survival | 2 years
  The number (%) of participants who do not show evidence of disease progression (according to RECIST criteria)at 2 years post initial administration of the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Martin E Guiterrez, MD, Principal Investigator — Holy Cross Hospital
Locations (1):
- Holy Cross Hospital, Inc, Fort Lauderdale, Florida, United States

REFERENCES:
- See also: Holy Cross Hospital — http://www.holy-cross.com/